CLINICAL TRIAL: NCT01317511
Title: Overnight Protein Supply as a Dietary Strategy to Improve Muscle Mass in Elderly.
Brief Title: Protein Supply in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. LJC van Loon, MaastrichtUMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 09-3-078.3
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Muscle Synthesis
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein (Experimental): Protein drink
  Interventions: Dietary Supplement: Protein
- Placebo (Placebo Comparator): water
  Interventions: Dietary Supplement: Protein

INTERVENTIONS:
Dietary Supplement: Protein — Protein drink
  Other Names: casein vs water

SUMMARY:
Stimulating overnight muscle protein synthesis, might augment muscle hypertrophy, increase mitochondrial mass, and/or improve muscle tissue repair. The goal of this proposal will be to provide further insight into the responsiveness of the muscle protein synthetic machinery to food intake in relation to age.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age between 65 and 80 years
* BMI < 30 kg/m2

Exclusion Criteria:

* Type 2 diabetic patients
* Use of medication
* All co morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. artrosis, arthritis, spasticity/rigidity, all neurological disorders and paralysis).
* Use of anticoagulants, blood diseases, allergy for lidocain.
* Contra indications for the use of a nasogastric tube: high risk of aspiration, gastric stasis, gastro-oesophageal reflux, upper gastrointestinal stricture, nasal injuries and base of skull fractures.
* Patients suffering from PKU (Phenylketonuria).

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Protein synthesis | overnight (12 h)
  Overnight protein synthesis

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Prof., Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356